CLINICAL TRIAL: NCT03815292
Title: Multicenter Double-blind Placebo-controlled Randomized Parallel-group Clinical Study of Efficacy and Safety of MMH-MAP in the Treatment of Mild Cognitive Impairment in Subjects in Early Rehabilitation Period of Ischemic Stroke
Brief Title: Clinical Trial of Efficacy and Safety of MMH-MAP in the Treatment of Mild Cognitive Impairment in Early Recovery Stage After Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-MAP-001
Record Dates: First submitted 2018-11-11; First posted 2019-01-24 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2019-08

CONDITIONS: Mild Cognitive Impairment; Ischemic Stroke
MeSH Terms: conditions — Cognitive Dysfunction; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMH-MAP (Experimental): Tablet for oral use. Dose per administration: 2 tablets. 2 tablets twice daily (4 tablets/day). The tablets should be held in mouth without chewing until complete dissolution. The duration of treatment will be 24 weeks.
  Interventions: Drug: MMH-MAP
- Placebo (Placebo Comparator): Placebo for 24 weeks, according to the MMH-MAP dosing regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MMH-MAP — Oral administration
  Arms: MMH-MAP
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is:

* to evaluate efficacy of MMH-MAP in the treatment of mild cognitive impairment in subjects in early rehabilitation period of ischemic stroke
* to evaluate safety of MMH-MAP in the treatment of mild cognitive impairment in subjects in early rehabilitation period of ischemic stroke

DETAILED DESCRIPTION:
A double-blind, placebo-controlled randomized clinical trial in parallel groups.

The study patients are subjects of either gender, aged 45-80 years old, after an ischemic stroke within 3-6 months prior to enrollment and confirmed by neuroimaging, having mild cognitive impairment.

After the patients provide signed Participant Information Sheet and Informed Consent, they will be interviewed for complaints and medical history and undergo physical examination and laboratory tests. The doctor will rate the severity of patients' cognitive impairments on the Mini Mental State Examination (MMSE) scale and Montreal Cognitive Assessment (MoCA) scale, assess their performance in activities of daily living on the Barthel Index scale [Collin C, Wade DT, Davies S, Horne V. "The Barthel ADL Index: a reliability study." Int Disability Study.1988;10:61-63.], and administer the Stroke Specific Quality of Life Scale (SS-QOL) questionnaire [Williams LS, Weinberger M, Harris LE, Clark DO, Biller J. Development of a stroke-specific quality of life scale. Stroke 1999 Jul;30(7):1362-9]. Eligible participants will have to have moderate cognitive impairments (MMSE score - at least 21 and MoCA - less than 26). Therapy received by patients for their co-morbidities and primary diagnosis will be recorded. All women of childbearing potential will be administered pregnancy tests.

If a patient meets all inclusion criteria and does not have any exclusion criteria at Visit 1, he/she is randomized to one of the two groups: group 1 will receive MMH-MAP at 2 tablets twice daily; group 2 will receive Placebo using the study product dosing regimen. The total duration of follow-up and treatment will be 28 weeks, which will include 5 additional visits.

At Visit 2 (Week 4±7 days), the doctor records patients' complaints and physical examination data, reviews the progress of study and basic and concomitant therapy, and assesses treatment safety and patient compliance with treatment.

At Visit 3 (Week 8±7 days), Visit 4 (Week 16±7 days), and Visit 5 (Week 24±7 days), the doctor assesses patients' cognitive impairments (MoCA) and performance in activities of daily living (the Barthel Index). The patients complete the SS-QOL questionnaire.

At Visit 5 (Week 24±7 days), the doctor will additionally complete the Clinical Global Impression Efficacy Index (CGI-EI) scale [Guy W, editor. ECDEU Assessment Manual for Psychopharmacology. 1976 Rockville, MD, U.S. Department of Health, Education, and Welfare] and collect samples for laboratory testing. The patient stops taking the study drug.

After four weeks following the end of study therapy patients complete a follow-up visit -Visit 6 (Week 28±7 days). The patients are interviewed for complaints and undergo physical examination, with a check on their concomitant and primary therapies as well as on the safety of study treatment. The doctor assesses patients' cognitive impairments (MoCA) and performance in activities of daily living (the Barthel Index) and administers the SS-QOL questionnaire.

The total length of the observation period will be 28 weeks. During the study, symptomatic therapy and therapy for underlying chronic conditions are allowed with the exception of the drugs indicated in the section "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex, aged 45 to 80 years old inclusively.
2. Patients with a history of one stroke sustained 3 to 6 months prior to study entry and confirmed by neuroimaging.
3. Patients with cognitive impairment (MoCA score < 26).
4. Patients with moderate performance in activities of daily living (Barthel score = 61-80).
5. Agreement to use a reliable method of birth control for the duration of the study (men and women of reproductive potential).
6. Availability of signed patient information sheet (Informed Consent form) for participation in the clinical trial.

Exclusion Criteria:

1. Patients with a history of subarachnoid/parenchymatous/ventricular hemorrhage, brain neoplasm, or any other condition which has caused neurological dysfunction.
2. History of central nervous system (CNS) disorders, including:

   * inflammatory diseases of the CNS (G00-G09)
   * systemic atrophies primarily affecting the CNS (G10-G13)
   * extrapyramidal and movement disorders (G20-G26)
   * other degenerative diseases of the nervous system (G30-G32)
   * demyelinating diseases of the CNS (G35-G37)
   * epilepsy (G40-41)
   * polyneuropathies and other disorders of the peripheral nervous system (G60-64), with marked movement and/or sensory impairments that cause movement disorders
   * diseases of neuromuscular junction and muscle (G70-73)
   * hydrocephalus (G91)
   * compression of brain (G93.5).
3. Dementia (20 or less on the MMSE score).
4. Speech disorders affecting investigator-patient communication.
5. Prior diagnosis of heart failure defined by the New York Heart Association classification (1964) as IV Functional Classification or poorly treated hypothyroidism or diabetes mellitus.
6. Patients having unstable angina or myocardial infarction in the past 6 months.
7. History/suspicion of oncology of any location (except for benign neoplasms).
8. Any other co-morbidity which, in the opinion of the investigator, may affect patient participation in the clinical trial.
9. Patients allergic to/intolerant of any components of the study treatment.
10. Patients with hereditary lactose intolerance.
11. Malabsorption syndrome, including congenital or acquired lactase deficiency (or any other disaccharidase deficiency) and galactosemia.
12. Pregnancy, breast-feeding or unwillingness to use birth control during the study.
13. Patients who, from the investigator's point of view, will not comply with the observation requirements of the study or adhere to study drug dosing regimens.
14. Patients with a history of non-adherence to medication; mental disorder (except for cognitive deficits); or alcoholism or abuse of psychoactive substances, which, in the investigator's opinion, will compromise compliance with study procedures.
15. Patients who have used medications listed in 'Prohibited Concomitant Treatment' in the past week.
16. Participation in other clinical trials in the previous 3 months.
17. Patients who are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
18. Patients who work for MATERIA MEDICA HOLDING (i.e. the company's employees, temporary contract workers, appointed officials responsible for carrying out the research or immediate relatives of the aforementioned).

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- Russia (28):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Belgorod Regional Clinical Hospital of St. Joseph, Belgorod
  - Non-State Healthcare Institution "Divisional Hospital at the Bryansk-2 station of the open joint-stock company Russian Railways", Bryansk
  - Bryansk Regional Hospital № 1, Bryansk
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University" of the Ministry of Healthcare of the Russian Federation, Kazan'
  - Scientific-Research Institute - Regional Clinical Hospital №1 named after Professor S.V. Ochapovsky, Krasnodar
  - The State Budget Health Care institution of Moscow the City "City clinical hospital No. 12 of the Administration of Health Care of Moscow City", Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow City Clinical Hospital No. 1 named after. N.I. Pirogov Moscow Department of Health, Moscow
  - City Clinical Hospital named after SI. Spasokokukotsky Department of Health of Moscow, Moscow
  - City Clinical Hospital №5 of Nizhny Novgorod region of Nizhny Novgorod, Nizhny Novgorod
  - Privolzhskiy Research Medical University, Nizhny Novgorod
  - State budgetary institution of public health services of the Nizhniy Novgorod region "Nizhegorod Regional Clinical Hospital named after NA Semashko", Nizhny Novgorod
  - Pyatigorsk City Clinical Hospital № 2, Pyatigorsk
  - Ryazan State Medical University named after academician I.P. Pavlov, Ryazan
  - St. Petersburg I. I. Dzhanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - State budgetary institution of health care of the Samara region "Samara City Clinical Hospital № 1 named after NI Pirogov", Samara
  - Republican Clinical Hospital №4, Saransk
  - Saratov State Medical University named after V. I. Razumovsky, Saratov
  - St. Petersburg State Budgetary Institution "City Hospital No. 40 in the Kurortny District", Sestroretsk
  - Smolensk State Medical University, Smolensk
  - State budgetary institution of health care of the Tver region "Regional Clinical Treatment and Rehabilitation Center", Tver'
  - State Healthcare Institution Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - State budgetary health care institution of the Vladimir region "Regional Clinical Hospital", Vladimir
  - Volgograd State Medical University, Volgograd
  - Voronezh Regional Clinical Hospital № 1, Voronezh
  - Vsevolozhsk Clinical Interdistrict Hospital, Vsevolozhsk
  - State Institution of Health of the Yaroslavl Region Clinical Hospital No. 8, Yaroslavl

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 276 patients signed informed consent. After screening procedures, data from 1 patient did not meet the inclusion / exclusion criteria. The study randomized 275 patients.
Period: Overall Study
Arm/Group | MMH-MAP | Placebo
Started | 135 | 140
Completed | 135 | 140
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMH-MAP | Placebo | Total
Number analyzed (Participants) | 135 | 140 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.7) | 63.5 (8.5) | 64.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 124
  Male | 73 | 78 | 151
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 135 | 140 | 275

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Improved Cognitive Function (The Montreal Cognitive Assessment Test Total Score of the Baseline +1 or More)
Description: MoCa is the test for assessment of cognitive impairment. The score ranges between 0 and 30. A score of 26-30 is normal. A score less than 26 is considered as mild cognitive impairment. Higher values represent a better outcome.
Time Frame: 24 weeks of the treatment as compared to the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 135 | 140
Participants | 124 | 115
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Test type: Superiority; p = 0.02, Fisher Exact

2. Other Pre Specified Outcome: Change in MoCA (The Montreal Cognitive Assessment Test) Score
Description: as for outcome 1
Time Frame: 24 weeks of the treatment as compared to the baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 135 | 140
score on a scale
  Baseline | 19.4 (2.3) | 19.2 (2.5)
  After 24 weeks | 23.3 (2.7) | 22.5 (3.0)
  ∆ between baseline and after 24 weeks | 3.8 (2.4) | 3.1 (2.9)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; This analysis applies to ∆ between baseline and after 24 weeks total scores row; Test type: Superiority; p = 0.0445, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Percentage of Patients With Improved Performance in Activities of Daily Living (Barthel Index Score of the Baseline + 5 or More)
Description: Scale for measurement of performance in activities of daily living (ADL).The maximum score is 100. A score of 91-99 stands for mild dependence in ADL performance, 61-90 - for moderate dependence in ADL performance, 21-60 - for severe dependence in ADL performance, 0-20 - for complete dependence in ADL performance. Higher values represent a better outcome.
Time Frame: 24 weeks of the treatment as compared to the baseline
Population: According to this criterion, data were obtained for 131 patients of the MMH-MAP group and 127 patients of the Placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 131 | 127
Participants | 118 | 102
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Test type: Superiority; p = 0.0345, Fisher Exact

4. Other Pre Specified Outcome: Change in Barthel Index Score
Description: as for outcome 3
Time Frame: 24 weeks of the treatment as compared to the baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 135 | 140
score on a scale
  Baseline | 74.7 (5.4) | 74.8 (5.7)
  After 24 weeks | 89.7 (8.7) | 86.6 (11.3)
  ∆ between baseline and after 24 weeks | 14.9 (8.8) | 12.2 (10.4)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; This analysis applies to ∆ between baseline and after 24 weeks total scores row; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Change in SS-QOL (Stroke Specific Quality of Life Scale) Total Score
Description: Scale for assessment of health-related quality of life. The scale consists of 49 items in the 12 domains. Each domain consists of 3 to 10 items that are averaged to generate an overall score. Total score minimum value is 1 and maximum value is 245. Higher values represent a better outcome.
Time Frame: 24 weeks of the treatment as compared to the baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 135 | 140
score on a scale
  Baseline | 155.6 (33.0) | 156.6 (32.6)
  After 24 weeks | 184.2 (35.3) | 173.7 (38.0)
  ∆ between baseline and after 24 weeks | 27.9 (26.1) | 17.5 (26.5)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; This analysis applies to ∆ between baseline and after 24 weeks total scores row; Test type: Superiority; p = 0.0016, t-test, 2 sided

6. Other Pre Specified Outcome: The CGI-EI (Clinical Global Impression Efficacy Index) Score
Description: Rating scale for assessment of the therapeutic effect of treatment and associated side effects. The scale consists of 2 items: therapeutic effect and side effects. Scores in therapeutic effect range from 1 (marked improvement) to 13 (unchanged or worse). Scores in side effects range from 0 (no side effects) to 3 (side effects outweigh therapeutic effects). Efficacy index ranges between 0 and 16. Higher values represent a worse result.
Time Frame: 24 weeks of the treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 131 | 127
score on a scale
  Therapeutic effect | 5.7 (3.3) | 6.9 (3.4)
  Side effects | 0.1 (0.4) | 0.1 (0.4)
  Efficacy index | 5.8 (3.4) | 7.0 (3.4)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; This analysis applies to Therapeutic effect row; Test type: Superiority; p = 0.0054, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: MMH-MAP vs Placebo; This analysis applies to Side effects row; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: MMH-MAP vs Placebo; This analysis applies to Efficiency index row; Test type: Superiority; p = 0.0042, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Change in MoCA (The Montreal Cognitive Assessment Test) Score During Follow-up
Description: Test for assessment of cognitive impairment. The score ranges between 0 and 30. A score of 26-30 is normal. A score less than 26 is considered as mild cognitive impairment. Higher values represent a better outcome.
Time Frame: 24 and 28 weeks of the study
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 131 | 127
score on a scale
  After 24 weeks | 23.3 (2.7) | 22.5 (3.0)
  After 28 weeks | 23.6 (3.1) | 22.7 (3.1)
  ∆ between 24 and 28 weeks | 0.4 (1.3) | 0.3 (1.4)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; This analysis applies to ∆ between 24 and 28 weeks total scores row; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney)

8. Other Pre Specified Outcome: Change in Barthel Index Score During Follow-up
Description: Scale for measurement of performance in activities of daily living (ADL). The maximum score is 100. A score of 91-99 stands for mild dependence in ADL performance, 61-90 - for moderate dependence in ADL performance, 21-60 - for severe dependence in ADL performance, 0-20 - for complete dependence in ADL performance. Higher values represent a better outcome.
Time Frame: 24 and 28 weeks of the study
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 131 | 127
score on a scale
  After 24 weeks | 89.7 (8.7) | 86.6 (11.3)
  After 28 weeks | 90.6 (10.9) | 87.4 (10.1)
  ∆ between 24 and 28 weeks | 1.5 (3.1) | 0.6 (3.1)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; This analysis applies to ∆ between 24 and 28 weeks total scores row; Test type: Superiority; p = 0.0118, Wilcoxon (Mann-Whitney)

9. Other Pre Specified Outcome: Change in Total SS-QOL (Stroke Specific Quality of Life Scale) Score During Follow-up
Description: Scale for assessment of health-related quality of life. The scale consists of 49 items in the 12 domains.Each domain consists of 3 to 10 items that are averaged to generate an overall score.Total score minimum value is 1 and maximum value is 245.Higher values represent a better outcome.
Time Frame: 24 and 28 weeks of the study
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 131 | 127
score on a scale
  After 24 weeks | 184.2 (35.3) | 173.7 (38.0)
  After 28 weeks | 187.8 (37.7) | 174.7 (38.0)
  ∆ between 24 and 28 weeks | 4.1 (9.5) | 2.8 (10.2)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; This analysis applies to ∆ between 24 and 28 weeks total scores row; Test type: Superiority; p = 0.058, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the study - 28 weeks.
Arm/Group | MMH-MAP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/135 | 1/140
Serious Adverse Events (participants affected / at risk) | 4/135 | 3/140
Other Adverse Events (participants affected / at risk) | 37/135 | 39/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMH-MAP (N=135) | Placebo (N=140)
Limb vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) — Lower limb vein phlebothrombosis
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) — Deep vein thrombosis of the right leg
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) — Recurrent cerebral infarction
Nosocomial pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Early nosocomial right-sided mid-lobe pneumonia
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Acute abdomen
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 1 (1) — Repeated ischemic stroke in the vertebrobasilar basin with infarction in the left cerebellar hemisphere
Acute coronary syndrome (General disorders) | 0 (0) | 1 (1)
Recurrent stroke (Nervous system disorders) | 0 (0) | 1 (1) — Recurrent cryptogenic ischemic stroke in the vertebrobasilar basin
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMH-MAP (N=135) | Placebo (N=140)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in the upper abdomen (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 7 (7)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) — Upper lip herpes
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Itchy rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Limb pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive impairment (Nervous system disorders) | 1 (1) | 0 (0)
Memory disorder (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Heartbeat (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Protein in urine (Investigations) | 0 (0) | 2 (2)
Oxalates in urine (Investigations) | 1 (1) | 0 (0)
Abnormal urine test results (Investigations) | 0 (0) | 1 (1) — Leukocyte esterase, hemoglobin traces, nitrites, leukocytes, erythrocytes, bacteria in a small amount
Increased blood pressure (Investigations) | 0 (0) | 1 (1)
Increased liver enzyme levels (Investigations) | 0 (0) | 1 (1)
Blood pressure decrease (Investigations) | 1 (1) | 0 (0) — Decrease in blood pressure on an outpatient basis
Weight gain (Investigations) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (3) | 0 (0)
Hunger (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Affective lability (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Increased libido (Psychiatric disorders) | 1 (1) | 0 (0)
Low mood (Psychiatric disorders) | 0 (0) | 1 (1)
Sense of anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Hematoma due to trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT03815292/Prot_SAP_000.pdf